CLINICAL TRIAL: NCT07132268
Title: Using Diaphragmatic Ultrasound to Predict Acute Respiratory Distress (ARD) in Patients Aged 75 and Over Admitted to the Emergency Department for Acute Dyspnea : Prospective Multicenter Study.
Brief Title: Diaphragm Response in Elderly for Acute Monitoring
Acronym: DREAM
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier de Bethune (Network)
Responsible Party: Sponsor
Other Study IDs: 2025-01; ID-RCB (Other: 2025-A00728-41)
Record Dates: First submitted 2025-07-03; First posted 2025-08-20 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2026-01

CONDITIONS: Acute Dyspnea; Acute Respiratory Failure; Diaphragmatic Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute dyspnea is a common cause of emergency department admissions among elderly patients. Acute respiratory failure is often multifactorial and requires rapid and reliable evaluation. Currently, management relies on clinical, biological, and radiological assessments, but diaphragmatic ultrasound could provide an additional tool for real-time respiratory function evaluation. This study aims to integrate this non-invasive technology into the initial assessment of patients to improve care pathways. Hypothesis : Diaphragmatic ultrasound enables reliable assessment of respiratory function and can predict the need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 75 years
* Emergency admission for acute dyspnea
* Requiring an emergency ultrsoung.

Exclusion Criteria:

* Acute respiratory distress requiring immediate invasive or non-invasive ventilation
* Respiratory rate ≥ 25 breaths/min, and/or SpO2 ≤ 90% on room air, and/or PaO2 ≤ 60 mmHg
* Known diaphragmatic paralysis
* Patients with degenerative neuromuscular disease
* State of shock: systolic blood pressure < 90 mmHg and/or mean arterial pressure < 65 mmHg and/or presence of skin mottling and/or CTR > 3s
* Lactate levels > 2 mmol/L
* Hypercapnic respiratory acidosis (pH < 7.38 and PaCO2 > 45 mmHg)
* Dyspnea due to metabolic acidosis (e.g., diabetic ketoacidosis, renal failure)
* Dyspnea of traumatic origin
* Refusal to participate or inability to provide informed consent
* Patients deprived of liberty
* Patients under guardianship or curatorship

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients Aged 75 and Over Admitted to the Emergency Department for Acute Dyspnea
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Occurrence of a severe acute respiratory event within 7 days of admission | WITHIN 7 DAYS OF ADMISSION
  * Placement on invasive mechanical ventilation (intubation) or non invasive ventilation (NIV, high-flow oxygen therapy),
  * Respiratory death, confirmed by an independent adjudication committee blinded to the ultrasound results.
  Explanatory variable: The presence of impaired diaphragmatic function at admission will be defined by:
  * a Tdi (tele-inspiratory thickness) <10%, and/or
  * a diaphragmatic excursion <10 mm.

SECONDARY OUTCOMES:
Measurement of diaphragmatic excursion AND Etiology of acute dyspnea | within 7 days
  To study the association between diaphragmatic excursion curve parameters (EDR, inspiratory time, expiratory time, etc.) and the etiology of acute dyspnea in patients aged 75 years and older admitted for acute dyspnea
To evaluate the contribution of diaphragmatic ultrasound to the NEWS2 score performed on admission in predicting the occurrence of acute respiratory distress within 7 days. | within 7 days
  The discriminatory power of the NEWS2 score in predicting the occurrence of acute respiratory distress, the discriminatory power of the NEWS2 score combined with impaired diaphragmatic function on admission ultrasound.
  NEWS 2 : The higher the score, the greater the risk of clinical deterioration. 0-4 : low risk Score of 3 in any individual parameter : low-medium 5-6 : moderate risk
  > or = 7 : high risk

CONTACTS AND LOCATIONS:
Overall Officials: Alain-Eric DUBART, Study Director — Centre Hospitalier de Béthune-Beuvry
Locations (9):
- France (9):
  - Centre Hospitalier Victor Dupouy, Argenteuil
  - Centre Hospitalier de Béthune, Béthune
  - Centre Hospitalier de Douai, Douai
  - Centre Hospitalier Emile Roux, Le Puy-en-Velay
  - Centre Hospitalier Sud Ile-de-France, Melun
  - Centre Hospitalier de Roubaix, Roubaix
  - Centre Hospitalier de Saint-Lô, Saint-Lô
  - Centre Hospitalier de Tourcoing, Tourcoing
  - Centre Hospitalier de Valenciennes, Valenciennes